CLINICAL TRIAL: NCT01960075
Title: A Multicenter, Randomized, Blinded, Comparative Effectiveness Study of Fosphenytoin, Valproic Acid, or Levetiracetam in the Emergency Department Treatment of Patients With Benzodiazepine-refractory Status Epilepticus.
Brief Title: Established Status Epilepticus Treatment Trial
Acronym: ESETT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Michigan (Other); Medical University of South Carolina (Other); Children's National Research Institute (Other); University of Minnesota (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jaideep Kapur, MD, Professor of Neurology and Neuroscience, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18078; 119756 (Other: ClinicalTrials.gov); U01NS088034 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Benzodiazepine Refractory Status Epilepticus
Keywords: status epilepticus, refractory, benzodiazepine, fosphenytoin, levetiracetam, valproic acid
MeSH Terms: conditions — Status Epilepticus | interventions — fosphenytoin; Levetiracetam; Valproic Acid

STUDY DESIGN:
Intervention Model Description: ESETT had 478 enrollments. They were 16 re-enrollers. This was an EFIC trial so all consents happened after treatment and all enrollments went through the same process of consent even if they were re-enrolled. Some information presented here only includes the first 400 patients since there was a prespecified stopping rule and the trial stopped early for futility.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fosphenytoin (FOS) (Active Comparator): Administer 20 mg/Kg fosphenytoin intravenously up to a maximum dose of 1500 mg ( 75 Kg) over 10 minutes. Those weighing more than 75 Kg receive a fixed dose of 1500 fosphenytoin over 10 minutes.
  Interventions: Drug: Fosphenytoin
- Valproic acid (Active Comparator): Administer 40 mg/Kg valproic acid intravenously up to a maximum dose of 3000 mg (75 Kg) over 10 minutes. Those weighing more than 75 Kg receive a fixed dose of 3000 valproic acidover 10 minutes.
  Interventions: Drug: Valproic acid
- Levetiracetam (Active Comparator): Administer 60 mg/Kg levetiracetam intravenously up to a maximum dose of 4500 mg ( 75 Kg) over 10 minutes. Those weighing more than 75 Kg receive a fixed dose of 4500 levetiracetam over 10 minutes.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Fosphenytoin
  Arms: Fosphenytoin (FOS)
Drug: Levetiracetam
  Arms: Levetiracetam
Drug: Valproic acid
  Arms: Valproic acid

SUMMARY:
The primary objective is to determine the most effective and/or the least effective treatment of benzodiazepine-refractory status epilepticus (SE) among patients older than 2 years. There are three active treatment arms being compared: fosphenytoin (FOS),levetiracetam (LEV), and valproic acid (VPA).

The second objective is comparison of three drugs with respect to secondary outcomes.

The final objective is to ensure that the trial is informative for treatment of established SE in children by describing the effectiveness, safety, and rate of adverse reactions of these drugs in children.

ELIGIBILITY:
Inclusion Criteria: Patient witnessed to seize for greater than 5 minute duration prior to treatment with study drug; Patient received adequate dose of benzodiazepines. The last dose of a benzo was administered in the 5-30 minutes prior to study drug administration. The doses may be divided.; continued or recurring seizure in the Emergency Department; Age 2 years or older

Exclusion Criteria:Known pregnancy; Prisoner; Opt-out identification; Treatment with a second line anticonvulsant (FOS, PHT, VPA, LEV, phenobarbital or other agents defined in the MoP) for this episode of SE; Treatment with sedatives with anticonvulsant properties other than benzodiazepines (propofol, etomidate, ketamine or other agents defined in the MoP); Endotracheal intubation; Acute traumatic brain injury; Known metabolic disorder; Known liver disease; Known severe renal impairment; Known allergy or other known contraindication to FOS, PHT, LEV, or VPA; Hypoglycemia < 50 mg/dL; Hyperglycemia > 400 mg/dL; Cardiac arrest and post-anoxic seizures

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2015-10; Primary Completion 2019-02 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Kapur, MBBS, PhD, Study Chair — University of Virginia; Robert Silbergleit, MD, Principal Investigator — University of Michigan; James Chamberlain, MD, Principal Investigator — Children's National Research Institute; Jordan Elm, PhD, Principal Investigator — Medical University of South Carolina
Locations (65):
- United States (65):
  - Banner University Medical Center - South Campus, Tucson, Arizona
  - Banner University Medical Center-Tucson Campus, Tucson, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Davis Children's Hospital, Sacramento, California
  - San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Christiana Hospital, Newark, Delaware
  - A.I.DuPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - NYP Columbia University Medical Center, New York, New York
  - NYP Morgan Stanley Children's Hospital, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Crozer-Chester Medical Center, Chester, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital Episcopal Campus, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh UPMC, Pittsburgh, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Children's Medical Center UTSW, Dallas, Texas
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - Memorial Hermann Texas medical Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - University Health System University Hospital, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Background] Bleck T, Cock H, Chamberlain J, Cloyd J, Connor J, Elm J, Fountain N, Jones E, Lowenstein D, Shinnar S, Silbergleit R, Treiman D, Trinka E, Kapur J. The established status epilepticus trial 2013. Epilepsia. 2013 Sep;54 Suppl 6(0 6):89-92. doi: 10.1111/epi.12288. PMID 24001084
- [Background] Cock HR; ESETT Group. Established status epilepticus treatment trial (ESETT). Epilepsia. 2011 Oct;52 Suppl 8:50-2. doi: 10.1111/j.1528-1167.2011.03237.x. PMID 21967363
- [Derived] Coralic Z, Kapur J, Olson KR, Chamberlain JM, Overbeek D, Silbergleit R. Treatment of Toxin-Related Status Epilepticus With Levetiracetam, Fosphenytoin, or Valproate in Patients Enrolled in the Established Status Epilepticus Treatment Trial. Ann Emerg Med. 2022 Sep;80(3):194-202. doi: 10.1016/j.annemergmed.2022.04.020. Epub 2022 Jun 17. PMID 35718575
- [Derived] Rosenthal ES, Elm JJ, Ingles J, Rogers AJ, Terndrup TE, Holsti M, Thomas DG, Babcock L, Okada PJ, Lipsky RH, Miller JB, Hickey RW, Barra ME, Bleck TP, Cloyd JC, Silbergleit R, Lowenstein DH, Coles LD, Kapur J, Shinnar S, Chamberlain JM; Established Status Epilepticus Treatment Trial Study Group. Early Neurologic Recovery, Practice Pattern Variation, and the Risk of Endotracheal Intubation Following Established Status Epilepticus. Neurology. 2021 May 11;96(19):e2372-e2386. doi: 10.1212/WNL.0000000000011879. Epub 2021 Mar 23. PMID 34032604
- [Derived] Sathe AG, Brundage RC, Ivaturi V, Cloyd JC, Chamberlain JM, Elm JJ, Silbergleit R, Kapur J, Coles LD. A pharmacokinetic simulation study to assess the performance of a sparse blood sampling approach to quantify early drug exposure. Clin Transl Sci. 2021 Jul;14(4):1444-1451. doi: 10.1111/cts.13004. Epub 2021 May 1. PMID 33742783
- [Derived] Sathe AG, Underwood E, Coles LD, Elm JJ, Silbergleit R, Chamberlain JM, Kapur J, Cock HR, Fountain NB, Shinnar S, Lowenstein DH, Rosenthal ES, Conwit RA, Bleck TP, Cloyd JC. Patterns of benzodiazepine underdosing in the Established Status Epilepticus Treatment Trial. Epilepsia. 2021 Mar;62(3):795-806. doi: 10.1111/epi.16825. Epub 2021 Feb 10. PMID 33567109
- [Derived] Sathe AG, Mishra U, Ivaturi V, Brundage RC, Cloyd JC, Elm JJ, Chamberlain JM, Silbergleit R, Kapur J, Lowenstein DH, Shinnar S, Cock HR, Fountain NB, Babcock L, Coles LD. Early Exposure of Fosphenytoin, Levetiracetam, and Valproic Acid After High-Dose Intravenous Administration in Young Children With Benzodiazepine-Refractory Status Epilepticus. J Clin Pharmacol. 2021 Jun;61(6):763-768. doi: 10.1002/jcph.1801. Epub 2021 Jan 12. PMID 33336359
- [Derived] Scicluna VM, Biros M, Harney DK, Jones EB, Mitchell AR, Pentz RD, Silbergleit R, Speight CD, Wright DW, Dickert NW. Patient and Surrogate Postenrollment Perspectives on Research Using the Exception From Informed Consent: An Integrated Survey. Ann Emerg Med. 2020 Sep;76(3):343-349. doi: 10.1016/j.annemergmed.2020.03.017. Epub 2020 May 21. PMID 32446674
- [Derived] Chamberlain JM, Kapur J, Shinnar S, Elm J, Holsti M, Babcock L, Rogers A, Barsan W, Cloyd J, Lowenstein D, Bleck TP, Conwit R, Meinzer C, Cock H, Fountain NB, Underwood E, Connor JT, Silbergleit R; Neurological Emergencies Treatment Trials; Pediatric Emergency Care Applied Research Network investigators. Efficacy of levetiracetam, fosphenytoin, and valproate for established status epilepticus by age group (ESETT): a double-blind, responsive-adaptive, randomised controlled trial. Lancet. 2020 Apr 11;395(10231):1217-1224. doi: 10.1016/S0140-6736(20)30611-5. Epub 2020 Mar 20. PMID 32203691
- [Derived] Kapur J, Elm J, Chamberlain JM, Barsan W, Cloyd J, Lowenstein D, Shinnar S, Conwit R, Meinzer C, Cock H, Fountain N, Connor JT, Silbergleit R; NETT and PECARN Investigators. Randomized Trial of Three Anticonvulsant Medications for Status Epilepticus. N Engl J Med. 2019 Nov 28;381(22):2103-2113. doi: 10.1056/NEJMoa1905795. PMID 31774955
- [Derived] Sathe AG, Tillman H, Coles LD, Elm JJ, Silbergleit R, Chamberlain J, Kapur J, Cock HR, Fountain NB, Shinnar S, Lowenstein DH, Conwit RA, Bleck TP, Cloyd JC. Underdosing of Benzodiazepines in Patients With Status Epilepticus Enrolled in Established Status Epilepticus Treatment Trial. Acad Emerg Med. 2019 Aug;26(8):940-943. doi: 10.1111/acem.13811. Epub 2019 Jul 18. No abstract available. PMID 31161706
- See also: ESETT Website — http://nett.umich.edu/clinical-trials/esett

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ESETT had a total of 478 enrollments. This number includes 16 re-enrollers. This was an EFIC trial so all consents happened after treatment. All enrollments went through the same process of consent even if they were reenrolled. The first 400 patients were used in several parts of analyses since the trial stopped early for futility (prespecified).
Groups:
- Fosphenytoin (FOS): Administer 20 mg/Kg fosphenytoin intravenously up to a maximum dose of 1500 mg ( 75 Kg) over 10 minutes. Those weighing more than 75 Kg receive a fixed dose of 1500 fosphenytoin over 10 minutes.
  Fosphenytoin
- Valproic Acid: Administer 40 mg/Kg valproic acid intravenously up to a maximum dose of 3000 mg (75 Kg) over 10 minutes. Those weighing more than 75 Kg receive a fixed dose of 3000 valproic acidover 10 minutes.
  Valproic acid
- Levetiracetam: Administer 60 mg/Kg levetiracetam intravenously up to a maximum dose of 4500 mg ( 75 Kg) over 10 minutes. Those weighing more than 75 Kg receive a fixed dose of 4500 levetiracetam over 10 minutes.
  Levetiracetam
Period: Overall Study
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Started | 149 | 149 | 180
Completed | 141 | 146 | 173
Not Completed | 8 | 3 | 7

BASELINE CHARACTERISTICS:
Population: The difference from Participant Flow is because the total of 384 is from the first 400 patients and excludes 16 re-enrollers in the study, and the first 400 patients were used because of the prespecified stopping rule and the trial stopped for futility.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam | Total
Number analyzed (Participants) | 118 | 121 | 145 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (25.4) | 32.2 (25.4) | 33.3 (26.0) | 32.8 (25.6)
Age, Customized [Count of Participants; unit: Participants]
  Age: 0 - 5 yr | 24 | 28 | 30 | 82
  Age: 6 - 10 yr | 15 | 7 | 17 | 39
  Age: 11 - 20 yr | 10 | 18 | 9 | 37
  Age: 21 - 40 yr | 20 | 19 | 31 | 70
  Age: 41 - 60 yr | 26 | 26 | 34 | 86
  Age: => 61 yr | 23 | 23 | 24 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 56 | 68 | 171
  Male | 71 | 65 | 77 | 213
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 49 | 54 | 62 | 165
  Race/Ethnicity: White | 49 | 49 | 62 | 160
  Race/Ethnicity: Other, >1 race, or unknown | 20 | 18 | 21 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Ethnicity | 18 | 22 | 23 | 63
Prior history of epilepsy [Count of Participants; unit: Participants] | 80 | 83 | 97 | 260
Final Diagnosis [Count of Participants; unit: Participants]
  Seizure/Status Epilepticus | 104 | 102 | 128 | 334
  Non-epileptic spell | 11 | 13 | 13 | 37
  Unable to adjudicate | 3 | 6 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Cessation of Status Epilepticus - Intention to Treat
Description: Determined by the absence of clinically apparent seizures and improving consciousness at 1 hour without other anticonvulsant medications. Intention to treat
Time Frame: Within 60 minutes after the start of study drug infusion
Population: The difference from Participant Flow is because the total of 384 is from the first 400 patients and excludes 16 re-enrollers in the study. The first 400 patients were used because of the prespecified stopping rule and the trial stopped for futility.
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 118 | 121 | 145
Participants | 53 | 56 | 68

2. Primary Outcome: Number of Participants With Clinical Cessation of Status Epilepticus - Per-protocol Analysis
Description: Determined by the absence of clinically apparent seizures and improving consciousness at 1 hour without other anticonvulsant medications. Per-protocol analysis
Time Frame: Within 60 minutes after the start of study drug infusion
Population: The analysis population for this outcome is the Per-protocol population, which is all patients who completed the study without major protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 79 | 91 | 109
Participants | 37 | 43 | 51

3. Primary Outcome: Number of Participants With Clinical Cessation of Status Epilepticus - Adjudicated Outcomes Analysis
Description: Determined by the absence of clinically apparent seizures and improving consciousness at 1 hour without other anticonvulsant medications. The Adjudicated outcomes analysis is different from Outcome measure 1 because a central clinical phenomenology core of four neurologists adjudicated from the medical records the time to seizure cessation, the time in status epilepticus before trial-drug initiation, and the cause of the seizure. For each enrollment, two neurologists from this core group conducted independent initial reviews and then determined a consensus or consulted a third adjudicator, as needed. Adjudicators were unaware of the treatment assignments and made determinations by medical record review.
Time Frame: Within 60 minutes after the start of study drug infusion
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 118 | 121 | 145
Participants | 57 | 60 | 67

4. Secondary Outcome: Number of Participants With Admission to Intensive Care Unit
Description: ICU admission is recorded as occurring only if the ICU is the initial inpatient unit for the patient.
Time Frame: Admission to intensive care unit after start of study drug infusion, where the ICU is the initial inpatient unit for the patient
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 118 | 121 | 145
Participants | 70 | 71 | 87

5. Secondary Outcome: Length of ICU Stay
Description: Length of stay is determined by the number of calendar days after the day of ED arrival until hospital discharge or subject end-of-study.
Time Frame: number of calendar days after the day of ED arrival until hospital discharge or subject end-of-study
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 118 | 121 | 145
days | 1 [0 to 3] | 1 [0 to 3] | 1 [0 to 3]

6. Secondary Outcome: Minutes From Start of Trial Drug Infusion to Termination of Seizures for Patients With Treatment Success
Description: The time to termination of seizures is the interval from the start of study drug infusion to cessation of clinically apparent seizure in those who meet the primary outcome.
Time Frame: start of drug infusion to seizure cessation
Population: The analysis population here is different than Participant Flow because it includes only the patients who had this data available. The first 400 patients were used because of the prespecified stopping rule and the trial stopped for futility.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 15 | 10 | 14
minutes | 11.7 [7.5 to 20.9] | 7.0 [4.6 to 14.9] | 10.5 [5.7 to 15.5]

7. Secondary Outcome: Number of Participants With Seizure Cessation Within 20 Minutes for Patients With Treatment Success
Description: Number of participants with seizure cessation within 20 minutes of study drug initiation for patients with treatment success. This outcome measure was only reported in the Supplementary materials to the Primary Paper.
Time Frame: within 20 minutes
Population: The population is different than Participant flow because it is only those with treatment success. This outcome measure was only reported in the Supplementary materials to the Primary Paper.
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 53 | 55 | 68
Participants | 43 | 43 | 53

8. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay in days
Time Frame: length of hospital stay
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 118 | 121 | 145
days | 3 [1 to 6] | 3 [2 to 6] | 3 [1 to 7]

9. Other Pre Specified Outcome: Number of Participants With Safety Outcome: Life Threatening Hypotension
Description: Life-threatening hypotension within 60 minutes of the start of study drug infusion
Time Frame: within 60 minutes of the start of study drug infusion
Population: The first 400 patients were analyzed for this outcome. The first 400 patients were used because of the prespecified stopping rule and the trial stopped for futility.
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 125 | 125 | 150
Participants | 4 | 2 | 1

10. Other Pre Specified Outcome: Number of Participants With Safety Outcome: Life-threatening Cardiac Arrhythmia
Description: Life-threatening cardiac arrhythmia within 60 minutes of the start of study drug infusion
Time Frame: within 60 minutes of the start of study drug infusion
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 125 | 125 | 150
Participants | 0 | 0 | 1

11. Other Pre Specified Outcome: Number of Participants With Safety Outcome: Endotracheal Intubation
Description: Endotracheal intubation within 60 minutes of start of study drug infusion
Time Frame: within 60 minutes of start of study drug infusion
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 125 | 125 | 150
Participants | 33 | 21 | 30

12. Other Pre Specified Outcome: Number of Participants With Safety Outcome: Acute Anaphylaxis
Description: Acute anaphylaxis is defined as a clinical presentation consistent with life threatening allergic reaction occurring within 6 hours of the start of study drug infusions and manifested as urticaria in combination with either (1) a systolic blood pressure of < 90 mmHg sustained for greater than 5 minutes, or (2) objective evidence of airway obstruction, and for which the patient was treated with antihistamines and/or steroids.
Time Frame: within 6 hours of the start of study drug infusions
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 125 | 125 | 150
Participants | 0 | 0 | 0

13. Other Pre Specified Outcome: Number of Participants With Safety Outcome: Acute Respiratory Depression
Description: Respiratory depression is defined as impairment of ventilation or oxygenation necessitating definitive endotracheal intubation and mechanical ventilation. It is distinct from intubations performed only for airway protection in those with decreased levels of consciousness. It does not include those getting only supraglottic airways or transient bag-valve-mask support.
Time Frame: 24 hours
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 125 | 125 | 150
Participants | 16 | 10 | 12

14. Other Pre Specified Outcome: Number of Participants With Safety Outcome: Hepatic Transaminase or Ammonia Elevations
Description: Safety outcome: Hepatic transaminase or ammonia elevations
Time Frame: 24 hours
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 125 | 125 | 150
Participants | 0 | 1 | 1

15. Other Pre Specified Outcome: Number of Participants With Safety Outcome: Purple Glove Syndrome
Description: Purple glove syndrome is defined as the presence of all three of the findings of the objective edema: discoloration, and pain in the distal extremity in which study drug was administered, with or without known extravasation, and for which there is no other evident etiology.
Time Frame: 24 hours
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 125 | 125 | 150
Participants | 0 | 0 | 0

16. Other Pre Specified Outcome: Number of Participants With Safety Outcome: Death
Description: Safety outcome: Death
Time Frame: 30 days
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 125 | 125 | 150
Participants | 3 | 2 | 7

17. Other Pre Specified Outcome: Number of Participants With Safety Outcome: Acute Seizure Recurrence
Description: acute seizure recurrence 60 minutes to 12 hours after start of study drug infusion
Time Frame: 60 minutes to 12 hours after start of study drug infusion
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
Number analyzed (Participants) | 125 | 125 | 150
Participants | 14 | 14 | 16

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected through the first 24 hours after enrollment, for the duration of the trial.
Description: All-Cause mortality data was collected for the first 400 subjects, which is why the numbers in the All-cause mortality section differ from Participant flow. The first 400 patients were used because of the prespecified stopping rule and the trial stopped for futility.
Arm/Group | Fosphenytoin (FOS) | Valproic Acid | Levetiracetam
All-Cause Mortality (participants affected / at risk) | 3/125 | 2/125 | 7/150
Serious Adverse Events (participants affected / at risk) | 57/125 | 46/125 | 64/150
Other Adverse Events (participants affected / at risk) | 28/125 | 22/125 | 25/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosphenytoin (FOS) (N=125) | Valproic Acid (N=125) | Levetiracetam (N=150)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular spasm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Convulsion (Nervous system disorders) | 25 (26) | 23 (23) | 30 (32)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 12 (12) | 9 (9) | 15 (15)
Device malfunction (General disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 7 (7) | 6 (6) | 4 (4)
Hypothermia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 4 (4)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 8 (8) | 10 (10)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosphenytoin (FOS) (N=125) | Valproic Acid (N=125) | Levetiracetam (N=150)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 3 (3) | 8 (8) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 7 (7) | 1 (1) | 4 (4)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Postictal paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 3 (3)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT01960075/Prot_SAP_000.pdf
  • Informed Consent Form (2015-01-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT01960075/ICF_001.pdf